CLINICAL TRIAL: NCT00662558
Title: A Six Week Double-Blind, Randomized, Multicenter Comparison Study Of The Analgesic Effectiveness Of Celecoxib 200 Mg BID Compared To Tramadol Hydrochloride 50 Mg QID In Subjects With Chronic Low Back Pain
Brief Title: A Six Week Study Of The Pain Relieving Effects Of Celecoxib 200 Mg Twice Daily Compared To Tramadol 50 Mg Four Times Daily In Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191338
Record Dates: First submitted 2007-12-06; First posted 2008-04-21 (Estimated); Results first posted 2009-11-23 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Celecoxib; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- celecoxib (Experimental)
  Interventions: Drug: celecoxib
- tramadol (Active Comparator)
  Interventions: Drug: tramadol HCL

INTERVENTIONS:
Drug: celecoxib — 200 mg capsules BID for 6 weeks
  Arms: celecoxib
Drug: tramadol HCL — 50 mg capsules QID for 6 weeks
  Arms: tramadol

SUMMARY:
To compare the analgesic effectiveness of celecoxib and tramadol in subjects with Chronic Low Back Pain measured by the Numerical Rating Scale (NRS-Pain) at Week 6

ELIGIBILITY:
Inclusion Criteria:

* The subject presents with duration of chronic low back pain of > 3 months requiring regular use of analgesics (> 4 days/week), except for acetaminophen which cannot have been the sole analgesic used

Exclusion Criteria:

* The subject has chronic low back pain, which is neurologic in etiology (i.e., radiculopathy, neuropathy, myelopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (52):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Wildomar, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Cos Cob, Connecticut
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Woodstock, Georgia
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New Windsor, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, North Charleston, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Grapevine, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Angelo, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Weber City, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191338&StudyName=A%20Six%20Week%20Study%20Of%20The%20Pain%20Relieving%20Effects%20Of%20Celecoxib%20200%20Mg%20Twice%20Daily%20Compared%20To%20Tramadol%2050%20Mg%20Four%20Times%20Daily%20In%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: 200 mg capsules two times a day (BID) for 6 weeks
- Tramadol HCL: 50 mg capsules four times a day (QID) for 6 weeks
Period: Overall Study
Arm/Group | Celecoxib | Tramadol HCL
Started | 398 | 404
Received Treatment | 396 | 396
Completed | 342 | 294
Not Completed | 56 | 110
Not completed — Adverse Event | 21 | 59
Not completed — Lack of Efficacy | 4 | 7
Not completed — Lost to Follow-up | 13 | 10
Not completed — Other | 9 | 14
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Randomized But Did Not Receive Treatment | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Tramadol HCL | Total
Number analyzed (Participants) | 396 | 396 | 792
Age, Customized [Number; unit: participants]
  18 to 44 years | 164 | 167 | 331
  45 to 64 years | 191 | 182 | 373
  > = 65 years | 41 | 47 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 213 | 450
  Male | 159 | 183 | 342

OUTCOME MEASURES:

1. Primary Outcome: Treatment Responders Based on the Numerical Rating Scale-Pain (NRS-Pain)
Description: A subject who met the following criteria was considered as a successful responder at Week 6: completed 6 weeks of treatment with study medication and had a 30% improvement from Baseline to Week 6/ET on the NRS-Pain. NRS-Pain scale assessed the severity of a subject's lower back pain on a scale of 0 (No pain) and 10 (Worst possible pain).
Time Frame: Week 6 or Early Termination (ET)
Population: Intent-to-treat = all subjects who were randomized and received at least one dose of study medication. Missing values were imputed using last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  Responders | 254 | 218
  Non-responders | 142 | 178
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; Test type: Non-Inferiority or Equivalence — Differences in treatment proportions and the 95% confidence interval (CI) around the difference were estimated by calculating the risk difference between the treatment arms using a generalized linear model with treatment and center as factors. A lower 95% CI for the risk difference greater than -0.10 would demonstrate that celecoxib 200 mg BID is not inferior to tramadol hydrochloride 50 mg QID; Risk Difference (RD) = 0.0910, 95% CI [0.0255 to 0.1565]
Statistical Analysis 2: Comparison: Celecoxib vs Tramadol HCL; If celecoxib 200 mg BID was found to be non-inferior to tramadol hydrochloride 50 mg QID then the second step was to test the superiority of celecoxib 200 mg BID over tramadol hydrochloride 50 mg QID using a two-sided test of proportions. Differences in proportions were tested using the General Association Test of the Cochran-Mantel-Haenszel (CMH) procedure stratified by center; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel

2. Secondary Outcome: Change From Baseline in Severity of Chronic Low Back Pain as Measured by NRS-Pain
Description: NRS-Pain scale assessed the severity of a subject's lower back pain on a scale of 0 (No pain) and 10 (Worst possible pain). NRS-Pain scale: Change = mean score at Week 6/ET minus mean score at Baseline.
Time Frame: Baseline, Week 6/ET
Population: ITT. Missing values were imputed by LOCF. Number of subjects with NRS-Pain scale scores at Baseline and Week 6/ET: celecoxib n=386, tramadol HCl n=385.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
scores on a scale | -3.38 (0.12) | -3.25 (0.13)
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; The change from Baseline was compared between the two treatment groups using analysis of covariance (ANCOVA), with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.234, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI [-0.53 to 0.13], Standard Error of Mean 0.17 — The mean difference reported is the least squares (LS) mean difference

3. Secondary Outcome: Change From Baseline in Severity of Low Back Pain as Measured by Visual Analogue Scale (VAS)
Description: VAS was a 100 millimeter (mm) scale that subjects used to assess the severity of their lower back pain. Based on the following question, "During the past day, how much back pain did you have?", the subject was instructed to place a vertical line on the VAS to indicate the magnitude of his/her lower back pain. 0 mm = no pain and 100 mm = worst possible pain. VAS: Change = mean score at Week 6/ET minus mean score at Baseline.
Time Frame: Baseline, Week 6/ET
Population: ITT. Missing values were imputed by LOCF. Number of subjects with VAS scores at Baseline and Week 6/ET: celecoxib n=386, tramadol HCl n=385.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
mm | -34.78 (1.33) | -34.27 (1.42)
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.595, ANCOVA; Mean Difference (Final Values) = -0.94, 95% CI [-4.39 to 2.52], Standard Error of Mean 1.76 — The mean difference reported is the LS mean difference

4. Secondary Outcome: Patient's Global Assessment of Disease Activity
Description: Number of subjects with a graded level of disease activity using the Patient's Global Assessment of Disease Activity 5-point scale (1=very good, 2=good, 3=fair, 4=poor, and 5=very poor). Subjects were classified as "Improved" if their assessment reduced at least 2 grades from baseline or if their assessment changed to Grade 1 (Very Good). Subjects were classified as "Worsened" if their assessment increased at least 2 grades from baseline or if their assessment changed to Grade 5 (Very Poor). Subjects were classified as "No Change" otherwise.
Time Frame: Week 6/ET
Population: ITT. Number of subjects with Patient's Global Assessment of Disease Activity scores at Week 6/ET: celecoxib n=375, tramadol HCl n=367.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  Improved | 108 | 107
  No Change | 264 | 259
  Worsened | 3 | 1
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; CMH tests using row mean score and adjusted for center was used to compare the two treatment groups; Test type: Superiority or Other; p = 0.829, Cochran-Mantel-Haenszel

5. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: Number of subjects with a physician's grading of disease activity using the Physician's Global Assessment of Disease Activity 5-point scale ((1=very good, 2=good, 3=fair, 4=poor, and 5=very poor). Subjects were classified as "Improved" if their assessment reduced at least 2 grades from baseline or if their assessment changed to Grade 1 (Very Good). Subjects were classified as "Worsened" if their assessment increased at least 2 grades from baseline or if their assessment changed to Grade 5 (Very Poor). Subjects were classified as "No Change" otherwise.
Time Frame: Week 6/ET
Population: ITT. Number of subjects with Physician's Global Assessment of Disease Activity scores at Week 6/ET: celecoxib n=368, tramadol HCl n=361.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  Improved | 113 | 102
  No Change | 253 | 258
  Worsened | 2 | 1
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; CMH tests using row mean score and adjusted for center was used to compare the two treatment groups; Test type: Superiority or Other; p = 0.470, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score
Description: Each subject assessed his/her own disability due to low back pain using the RMDQ worksheet, which consisted of 24 statements of disability. The RMDQ total score was calculated as the total number of statements that were checked; the RMDQ total scores could have ranged from 0 to 24, with higher scores indicating greater disability. RMDQ: Change = mean score at Week 6/ET minus mean score at Baseline.
Time Frame: Baseline, Week 6/ET
Population: ITT. Missing values were imputed by LOCF. Number of subjects with Roland-Morris Disability total scores at Baseline and Week 6/ET= celecoxib n=391, tramadol n=389.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
scores on a scale | -4.90 (0.26) | -4.45 (0.25)
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.339, ANCOVA; Mean Difference (Final Values) = -0.31, 95% CI [-0.95 to 0.33], Standard Error of Mean 0.32 — The mean difference reported is the LS mean difference

7. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory (m-BPI-sf)
Description: m-BPI-sf scale assessed pain severity (0 = no pain to 10 = worst possible pain), and pain interference of functional activities (0 = does not interfere to 10 = completely interferes) during the 24 hour follow-up period. Subjects indicated: how much pain now; worst pain; average level of pain; how much pain interfered with general activity, mood, walking ability, relations with other people, sleep, normal work (including housework), and enjoyment of life. m-BPI-sf: Change = mean score at Week 6/ET minus mean score at Baseline.
Time Frame: Baseline, Week 6/ET
Population: ITT. Missing values were imputed by LOCF. Number of subjects with m-BPI-sf scores at Baseline and Week 6/ET: celecoxib n=373, tramadol HCl n=367.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
scores on a scale
  How Much Pain Now | -2.87 (0.12) | -2.88 (0.13)
  Worst Pain in Past 24 Hours | -2.84 (0.13) | -2.87 (0.13)
  Average Pain in Past 24 Hours | -2.64 (0.11) | -2.59 (0.13)
  Pain Interfered With General Activity | -2.62 (0.12) | -2.57 (0.13)
  Pain Interfered With Mood | -2.38 (0.14) | -2.25 (0.15)
  Pain Interfered With Walking Activity | -2.26 (0.13) | -2.36 (0.13)
  Pain Interfered With Relations With Others | -1.79 (0.13) | -1.74 (0.14)
  Pain Interfered With Sleep | -2.52 (0.13) | -2.51 (0.15)
  Pain Interfered With Normal Work | -2.57 (0.13) | -2.46 (0.15)
  Pain Interfered With Enjoyment of Life | -2.43 (0.14) | -2.43 (0.15)
  Pain Interference Subscale | -2.37 (0.11) | -2.33 (0.12)
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; How Much Pain Now. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.741, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI [-0.36 to 0.25], Standard Error of Mean 0.16 — The mean difference reported is the LS mean difference
Statistical Analysis 2: Comparison: Celecoxib vs Tramadol HCL; Worst Pain in Past 24 Hours. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.796, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI [-0.38 to 0.29], Standard Error of Mean 0.17 — The mean difference reported is the LS mean difference
Statistical Analysis 3: Comparison: Celecoxib vs Tramadol HCL; Average Pain in Past 24 Hours. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.492, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI [-0.41 to 0.20], Standard Error of Mean 0.16 — The mean difference reported is the LS mean difference
Statistical Analysis 4: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With General Activity. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.893, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI [-0.28 to 0.33], Standard Error of Mean 0.16 — The mean difference reported is the LS mean difference
Statistical Analysis 5: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With Mood. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.618, ANCOVA; Mean Difference (Final Values) = -0.08, 95% CI [-0.40 to 0.24], Standard Error of Mean 0.16 — The mean difference reported is the LS mean difference
Statistical Analysis 6: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With Walking Activity. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.440, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI [-0.19 to 0.43], Standard Error of Mean 0.16 — The mean difference reported is the LS mean difference
Statistical Analysis 7: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With Relations With Others. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.806, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI [-0.25 to 0.32], Standard Error of Mean 0.14 — The mean difference reported is the LS mean difference
Statistical Analysis 8: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With Sleep. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.739, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI [-0.38 to 0.27], Standard Error of Mean 0.17 — The mean difference reported is the LS mean difference
Statistical Analysis 9: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With Normal Work. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.992, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.32 to 0.33], Standard Error of Mean 0.17 — The mean difference reported is the LS mean difference
Statistical Analysis 10: Comparison: Celecoxib vs Tramadol HCL; Pain Interfered With Enjoyment of Life. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.793, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI [-0.28 to 0.36], Standard Error of Mean 0.16 — The mean difference reported is the LS mean difference
Statistical Analysis 11: Comparison: Celecoxib vs Tramadol HCL; Pain Interference Subscale. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.973, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.27 to 0.28], Standard Error of Mean 0.14 — The mean difference reported is the LS mean difference

8. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale
Description: MOS sleep scale included the following attributes: sleep disturbance, snoring, awaken shortness of breath or headache, quantity of sleep, sleep adequacy, somnolence, Sleep Problem Index I, and Sleep Problem Index II. Score ranged from 0-100, with a higher score indicating more of the scale attribute (e.g., more sleep disturbance, etc.). A negative change indicated subject improvement. MOS sleep scale: Change = mean score at Week 6/ET minus mean score at Baseline.
Time Frame: Baseline, Week 6/ET
Population: ITT. Number of subjects with MOS scores at Baseline and Week 6/ET: n=celecoxib, tramadol HCl.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
scores on a scale
  Sleep Disturbance (n=374, 367) | -17.91 (1.23) | -16.34 (1.17)
  Snoring (n=372, 365) | -7.53 (1.31) | -5.10 (1.28)
  Awaken Shortness of Breath, Headache (n=374, 367) | -8.61 (1.27) | -6.21 (1.34)
  Quantity of Sleep (n=373, 365) | 0.00 (0.23) | 0.58 (0.28)
  Sleep Adequacy (n=373, 367) | 7.32 (1.48) | 9.67 (1.34)
  Somnolence (n=374, 366) | -9.63 (1.05) | -7.01 (1.16)
  Sleep Problem Index I (n=373, 367) | -11.59 (0.96) | -10.54 (0.92)
  Sleep Problem Index II (n=373, 367) | -12.97 (0.94) | -11.82 (0.89)
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; Sleep Disturbance. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.392, ANCOVA; Mean Difference (Final Values) = -1.29, 95% CI [-4.26 to 1.67], Standard Error of Mean 1.51 — The mean difference reported is the LS mean difference
Statistical Analysis 2: Comparison: Celecoxib vs Tramadol HCL; Snoring. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.691, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI [-3.94 to 2.61], Standard Error of Mean 1.67 — The mean difference reported is the LS mean difference
Statistical Analysis 3: Comparison: Celecoxib vs Tramadol HCL; Awaken Shortness of Breath or Headache. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.549, ANCOVA; Mean Difference (Final Values) = -0.87, 95% CI [-3.70 to 1.97], Standard Error of Mean 1.45 — The mean difference reported is the LS mean difference
Statistical Analysis 4: Comparison: Celecoxib vs Tramadol HCL; Quantity of Sleep. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.336, ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI [-0.67 to 0.23], Standard Error of Mean 0.23 — The mean difference reported is the LS mean difference
Statistical Analysis 5: Comparison: Celecoxib vs Tramadol HCL; Sleep Adequacy. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.370, ANCOVA; Mean Difference (Final Values) = -1.51, 95% CI [-4.83 to 1.80], Standard Error of Mean 1.69 — The mean difference reported is the LS mean difference
Statistical Analysis 6: Comparison: Celecoxib vs Tramadol HCL; Somnolence. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.341, ANCOVA; Mean Difference (Final Values) = -1.27, 95% CI [-3.90 to 1.35], Standard Error of Mean 1.34 — The mean difference reported is the LS mean difference
Statistical Analysis 7: Comparison: Celecoxib vs Tramadol HCL; Sleep Problem Index I. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.604, ANCOVA; Mean Difference (Final Values) = -0.59, 95% CI [-2.85 to 1.66], Standard Error of Mean 1.15 — The mean difference reported is the LS mean difference
Statistical Analysis 8: Comparison: Celecoxib vs Tramadol HCL; Sleep Problem Index II. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.547, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI [-2.92 to 1.55], Standard Error of Mean 1.14 — The mean difference reported is the LS mean difference

9. Secondary Outcome: Number of Subjects With Change From Baseline in MOS Optimal Sleep Scale Scores
Description: The Optimal Scale is scaled from 0 or 1 with 1 indicating 7 or 8 hours of sleep per night and 0 otherwise. Number of subjects with change of improvement (0 to 1), no change (1 to 1 or 0 to 0), or worsening (1 to 0) from baseline as indicated by the MOS Optimal sleep scale.
Time Frame: Baseline, Week 6/ET
Population: ITT. Number of subjects with MOS Optimal sleep scale scores at Week 6/ET: celecoxib n=373, tramadol HCl n=365.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  0 to 1 (Improvement) | 82 | 74
  1 to 1 (No change) | 94 | 70
  0 to 0 (No change) | 171 | 192
  1 to 0 (worsening) | 26 | 29
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; Optimal sleep was analyzed using CMH general association test; Test type: Superiority or Other; p = 0.196, Cochran-Mantel-Haenszel

10. Secondary Outcome: Change From Baseline in Work Limitations Questionnaire (WLQ)
Description: The WLQ included the following: Time Scale, Physical Scale, Output Scale, Mental-Interpersonal Scale, and Index Scale. The scales ranged from 0 (Limited none of the time) to 100 (Limited all of the time). A negative change indicated subject improvement.
Time Frame: Baseline, Week 6/ET
Population: ITT. Number of subjects with WLQ scores at Baseline and Week 6/ET: n=celecoxib, tramadol HCl.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
scores on a scale
  Time Scale (n=241, 239) | -11.55 (1.65) | -13.58 (1.52)
  Physical Scale (n=270, 254) | -13.68 (1.52) | -12.65 (1.45)
  Output Scale (n=256, 246) | -11.44 (1.54) | -11.69 (1.70)
  Mental-Interpersonal Scale (n=266, 252) | -9.06 (1.35) | -9.54 (1.51)
  Index Scale (n=223, 220) | -3.10 (0.36) | -3.14 (0.37)
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; Time Scale. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.252, ANCOVA; Mean Difference (Final Values) = 2.19, 95% CI [-1.56 to 5.94], Standard Error of Mean 1.91 — The mean difference reported is the LS mean difference
Statistical Analysis 2: Comparison: Celecoxib vs Tramadol HCL; Physical Scale. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.798, ANCOVA; Mean Difference (Final Values) = 0.48, 95% CI [-3.21 to 4.17], Standard Error of Mean 1.88 — The mean difference reported is the LS mean difference
Statistical Analysis 3: Comparison: Celecoxib vs Tramadol HCL; Output Scale. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.700, ANCOVA; Mean Difference (Final Values) = 0.74, 95% CI [-3.03 to 4.51], Standard Error of Mean 1.92 — The mean difference reported is the LS mean difference
Statistical Analysis 4: Comparison: Celecoxib vs Tramadol HCL; Mental-Interpersonal Scale. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.902, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI [-3.16 to 3.59], Standard Error of Mean 1.72 — The mean difference reported is the LS mean difference
Statistical Analysis 5: Comparison: Celecoxib vs Tramadol HCL; Index Scale. The change from Baseline was compared between the two treatment groups using ANCOVA, with treatment and center as factors, and Baseline value as a covariate; Test type: Superiority or Other; p = 0.581, ANCOVA; Mean Difference (Final Values) = 0.25, 95% CI [-0.65 to 1.16], Standard Error of Mean 0.46 — The mean difference reported is the LS mean difference

11. Secondary Outcome: Patient's Global Evaluation of Study Medication
Description: Number of subjects with an overall response to study medication of poor, fair, good, very good, and excellent.
Time Frame: Weeks 1, 3, and 6/ET
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  Week 1, Excellent | 46 | 38
  Week 1, Very Good | 97 | 83
  Week 1, Good | 126 | 137
  Week 1, Fair | 78 | 57
  Week 1, Poor | 23 | 18
  Week 3, Excellent | 52 | 41
  Week 3, Very Good | 104 | 97
  Week 3, Good | 122 | 105
  Week 3, Fair | 53 | 51
  Week 3, Poor | 23 | 14
  Week 6/ET, Excellent | 91 | 68
  Week 6/ET, Very Good | 123 | 112
  Week 6/ET, Good | 76 | 90
  Week 6/ET, Fair | 51 | 51
  Week 6/ET, Poor | 32 | 44
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; P-value reported is the overall p-value for Week 1; Test type: Superiority or Other; p = 0.614, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Celecoxib vs Tramadol HCL; P-value reported is the overall p-value for Week 3; Test type: Superiority or Other; p = 0.786, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Celecoxib vs Tramadol HCL; P-value reported is the overall p-value for Week 6/ET; Test type: Superiority or Other; p = 0.044, Cochran-Mantel-Haenszel

12. Secondary Outcome: Patient's Satisfaction Questionnaire (With Pain Relief Scale)
Description: Number of subjects at varying levels of pain relief (1 = very dissatisfied to 10 = very satisfied).
Time Frame: Week 6/ET
Population: ITT. Number of subjects with Patient's Satisfaction Questionnaire (with pain relief scale) scores at Week 6/ET: celecoxib n=373, tramadol HCl n=364.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  1 | 23 | 22
  2 | 15 | 18
  3 | 22 | 19
  4 | 22 | 20
  5 | 44 | 30
  6 | 23 | 29
  7 | 21 | 39
  8 | 63 | 56
  9 | 53 | 62
  10 | 87 | 69
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; CMH tests using row mean score and adjusted for center was used to compare the two treatment groups; Test type: Superiority or Other; p = 0.870, Cochran-Mantel-Haenszel

13. Secondary Outcome: Patient's Satisfaction Questionnaire (With Walking and Bending Ability Scale)
Description: Number of subjects at varying levels of pain relief (1 = very dissatisfied to 10 = very satisfied).
Time Frame: Week 6/ET
Population: ITT. Number of subjects with Patient's Satisfaction Questionnaire (with walking and bending ability scale) scores at Week 6/ET: celecoxib n=373, tramadol HCl n=364.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  1 | 24 | 15
  2 | 16 | 22
  3 | 19 | 20
  4 | 31 | 33
  5 | 35 | 40
  6 | 32 | 30
  7 | 35 | 37
  8 | 55 | 46
  9 | 56 | 77
  10 | 70 | 44
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; CMH tests using row mean score and adjusted for center was used to compare the two treatment groups; Test type: Superiority or Other; p = 0.545, Cochran-Mantel-Haenszel

14. Secondary Outcome: Chronic Low Back Pain Responders Based on VAS, Patient's Global, and RMDQ
Description: Subjects were successful responders if they had: > = 30% improvement from baseline to final visit in VAS assessment (as identified by 100 millimeter scale); > = 30% improvement from baseline to final visit in Patient's Global assessment (classified as improved if assessment reduced at least 2 grades from baseline or if assessment changed to Grade 1, worsened if assessment increased at least 2 grades from baseline or if assessment changed to Grade 5, or no change; and < 20% worsening from baseline to final visit in RMDQ assessment (lower scores indicated greater disability).
Time Frame: Week 6/ET
Population: ITT
Measure: Number; unit: participants
Arm/Group | Celecoxib | Tramadol HCL
Number analyzed (Participants) | 396 | 396
participants
  Responders | 213 | 196
  Non-responders | 183 | 200
Statistical Analysis 1: Comparison: Celecoxib vs Tramadol HCL; CMH test adjusted for center was used to compare the two treatment groups; Test type: Superiority or Other; p = 0.218, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | Celecoxib | Tramadol HCL
Serious Adverse Events (participants affected / at risk) | 1 | 0
Other Adverse Events (participants affected / at risk) | 89 | 171
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Celecoxib | Tramadol HCL
Coronary artery bypass (Surgical and medical procedures) | 1/396 | 0/396
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Celecoxib | Tramadol HCL
Constipation (Gastrointestinal disorders) | 8/396 | 25/396
Dry mouth (Gastrointestinal disorders) | 6/396 | 20/396
Nausea (Gastrointestinal disorders) | 31/396 | 70/396
Vomiting (Gastrointestinal disorders) | 5/396 | 28/396
Dizziness (Nervous system disorders) | 19/396 | 53/396
Headache (Nervous system disorders) | 41/396 | 54/396
Somnolence (Nervous system disorders) | 20/396 | 44/396
Pruritus (Skin and subcutaneous tissue disorders) | 2/396 | 23/396

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.